CLINICAL TRIAL: NCT06793904
Title: Comparative Study Between HOMA1-IR and HOMA2-IR in Prediction of Ovulation Outcome in Women With PCOS: A Prospective Cohort Study
Brief Title: Comparative Study Between HOMA1-IR and HOMA2-IR in Prediction of Ovulation Outcome in Women With PCOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N 364-2024; Cairo university (Other: Cairo university)
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Polycystic Ovarian Syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCOS (Experimental): Homeostatic model assessment for insulin resistance 1 will be calculated for all participants through the equation [glucose (mmol/L) × insulin (µU/L)]/22.5 while homeostatic model assessment for insulin resistance 2 will be calculated by the HOMA2 calculator. All women will be subjected to induction of ovulation using the Aromatase inhibitor Letrozole 2.5 mg tab twice daily from the 3rd day of the cycle for 5 days . Ultrasound follow up of follicular growth will be performed till dominant follicular size reaches 18-22 mm. FSH preparations were introduced as needed.
  Interventions: Drug: Aromatase inhibitor Letrozole

INTERVENTIONS:
Drug: Aromatase inhibitor Letrozole — 2.5 mg tab twice daily from the 3rd day of the cycle for 5 days

SUMMARY:
122 women diagnosed with PCOS seeking fertility in the fertility clinic at kasr Alainy hospital will be subjected to Homeostatic model assessment for insulin resistance 1 was calculated for all participants through the equation [glucose (mmol/L) × insulin (µU/L)]/22.5 while homeostatic model assessment for insulin resistance 2 was calculated by the HOMA2 calculator. All women will be subjected to induction of ovulation using the Aromatase inhibitor Letrozole 2.5 mg tab twice daily from the 3rd day of the cycle for 5 days . Ultrasound follow up of follicular growth will be performed till dominant follicular size reaches 18-22 mm. FSH preparations will be introduced as needed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* duration of infertility 1-4 years
* PCOS

Exclusion Criteria:

women with other causes of infertility (tubal factor assessed by laparoscopy or hysterosalpingogram, uterine cavity abnormality assessed by ultrasound or hysteroscopy or male factor assessed by seme analysis),

* endometriosis,
* ovarian cysts,
* endocrinological abnormalities (Diabetes mellitus, hypothalamic, pituitary or thyroid disorders, or hyperprolactinemia),
* women with history of poor ovarian response or ovarian hyperstimulation
* women with chronic diseases, chromosomal, autoimmune or coagulation defects, abnormal leucocytic count or other inflammatory markers
* Women with contraindications to pregnancy.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women diagnosed with PCOS
Enrollment: 122 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with successful ovulation | 5 days after treatment
  the dominant follicle reached 18 or more mm

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
upon reasonable request